CLINICAL TRIAL: NCT03255486
Title: Identification and Evaluation of Biomarkers of Resistance to Neoadjuvant Chemotherapy and Establishment of Preclinical Models of Resistance in Locally Advanced Breast Cancer
Brief Title: Identification and Evaluation of Biomarkers of Resistance to Neoadjuvant Chemotherapy (IDEA SEIN)
Acronym: IDEASEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICM2013/12
Record Dates: First submitted 2017-08-10; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood sample (Experimental): Blood samples will be taken by venipuncture during the initial assessment (4 tubes of 5 ml at diagnosis and 3 tubes of 5 ml to the following) These blood tests will be repeated after the first course, at the end of neoadjuvant chemotherapy and after surgery and will be carried out jointly to levies motivated by the balance sheet or the treatment of CS to avoid additional puncture.
  These samples will allow us to study the profiles of circulating tumor DNA, and miRNA tumor proteins (proteomics study).
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood samples will be taken by venipuncture during the initial assessment (4 tubes of 5 ml at diagnosis and 3 tubes of 5 ml to the following) These blood tests will be repeated after the first course, at the end of neoadjuvant chemotherapy and after surgery and will be carried out jointly to levies motivated by the balance sheet or the treatment of CS to avoid additional puncture.
  These samples will allow us to study the profiles of circulating tumor DNA, and miRNA tumor proteins (proteomics study).

SUMMARY:
Biomarkers of resistance to neoadjuvant chemotherapy in locally advanced breast cancer

DETAILED DESCRIPTION:
Identification and evaluation of biomarkers of resistance to neoadjuvant chemotherapy and establishment of preclinical models of resistance in locally advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

* proven invasive breast adenocarcinoma (cytology and / or biopsy).

  * locally advanced stage (tumor size greater than 2 cm).
  * neoadjuvant chemotherapy indication validated RCP
  * Patient eligible for neoadjuvant chemotherapy.
  * Performance Index according to WHO or less 1.
  * Patient aged 18 years and older.
  * Being affiliated to a social security scheme or an equivalent scheme of social protection
  * Obtaining signed informed consent, and that before any specific prequalification testing.

Exclusion Criteria:

* presence of metastatic disease at diagnosis.

  * Breast Cancer inflammatory.
  * rare histologic subtypes (non ductal lobular and not).
  * Other cancer (except basal cell skin carcinoma and cancer of the cervix in situ adequately treated and curative) treated in the previous 5 years.
  * Patient pregnant or nursing or of childbearing age without effective contraception.
  * Breast cancer in men.
  * legal incapacity or limited legal capacity. medical or psychological conditions allowing the subject to complete the study or to sign the consent (art. L.1121-6, L.1121-7, L.1211-8, L1211-9).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
predictive molecular abnormalities assessment | up to 5 years
  Highlighting and study of predictive molecular abnormalities of resistance to neoadjuvant chemotherapy in locally advanced breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ychou, Study Director — Institut régional du Cancer de Montpellier
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No